CLINICAL TRIAL: NCT04734301
Title: Efficacy of Intravaginal Electrical Stimulation With Different Treatment Frequency in Women With Idiopathic Overactive Bladder: A Prospective Randomized Controlled Trial
Brief Title: Intravaginal Electrical Stimulation With Different Treatment Frequency in Women With Idiopathic Overactive Bladder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Necmettin Yildiz, Clinical Professor, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-60116787-020-4274
Record Dates: First submitted 2021-01-25; First posted 2021-02-02 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Overactive Bladder
Keywords: idiopathic overactive bladder; intravaginal electrical stimulation; bladder training
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: IVES (2 times in a week) (Active Comparator): This group included the IVES in addition to all components of the BT. IVES was performed in lithotomy position via electrical stimulation device with a vaginal probe.
  Interventions: Device: Intravaginal Electrical Stimulation (2 times/week)
- Group 2: IVES (5 times in a week) (Experimental): This group also included the IVES in addition to all components of the BT as in Group 1. IVES performed in the same way as Group 1, except for frequency of treatment.
  Interventions: Device: Intravaginal Electrical Stimulation (5 times/week)

INTERVENTIONS:
Device: Intravaginal Electrical Stimulation (2 times/week) — IVES sessions were performed two times in a week, for 10 weeks. Every session lasted 20 minutes. The intervention comprised a 20-sessions treatment program of ES. The stimulation parameters were frequency at 10 Hz, a 5-10s work-rest cycle and 100 ms pulse width. The symmetric biphasic pulse wave could be delivered over a range of 0-100 mA. The intensity was controlled according to patients' discomfort level feedback.
  Arms: Group 1: IVES (2 times in a week)
Device: Intravaginal Electrical Stimulation (5 times/week) — IVES performed in the same way as Group 1, except for frequency of treatment. IVES sessions were performed five times in a week, for 4 weeks. Every session lasted 20 minutes. The intervention comprised a 20-sessions treatment program of ES. Stimulation parameters were the same as Group 1.
  Arms: Group 2: IVES (5 times in a week)

SUMMARY:
Electrical stimulation (ES) is one of the techniques used in urogynecological physiotherapy, which uses implanted or non-implanted electrodes. Intravaginal ES (IVES) is a conservative treatment option, described more than 40 years ago. IVES is used in patients with OAB and urge urinary incontinence (UUI), for detrusor inhibition. It has been suggested that IVES probably targets the detrusor muscle or pelvic floor muscle (PFM) or afferent innervation in UUI. According to the European Association Urology (EAU) Guidelines; in adults with urinary incontinence, ES may improve urinary incontinence compared to sham treatment. The IVES programs lasted between 4 weeks and 6 months in women with idiopathic OAB, although generally IVES was applied for 4-12 weeks. In most studies, IVES was applied 2-3 times a week, whereas in fewer studies it was applied more frequently. Despite that, no randomised studies compared different treatment frequencies in women with idiopathic OAB and thus, there is no evidence of which frequencies of treatment are the most effective ones. It should be kept in mind that different stimulation frequency may lead to different results. In addition, in the light of scientific evidence and our clinical experience, we think that this issue is still open for research. Better methodological quality studies are needed to obtain a higher level of scientific evidence and to know the optimal treatment frequency for OAB.

Our study is the first prospective randomized controlled trial that compares the efficacy of IVES with different treatment frequency in women with idiopathic OAB. In this study, we aimed to assess the efficacy of 2 times and 5 times in a week IVES added to BT on quality of life (QoL) and clinical parameters asssociated with idiopathic OAB. The results of the our study will be of great benefit in deciding or preferring the treatment frequency and total treatment duration of IVES for the women with idiopathic OAB and their physicians.

DETAILED DESCRIPTION:
This study is a prospective, randomized controlled trial. The trial is held at Urogynecological Rehabilitation Unit of Physical Medicine and Rehabilitation Department between February 2021 and July 2021. The local ethics committee approve the study (E-60116787-020-4274). All women are informed about the purpose and contents of the study and all women written consent to participate in the study.

A random allocation sequence was generated at 1:1 ratio. By using a random number generator, women are randomized into two groups as follows: Group 1 receive BT+IVES (2 times/week), Group 2 receive BT+IVES (5 times/week).

All women which are planned to treat during 20 sessions are included in this study.

Bladder Training (BT) All women were informed about BT for 30 minutes in two groups. Then it was given as a written brochure to be implemented as a home program. BT, consisting of four stages, did not contain any PFM training programs. At the first stage, all of the women visited the physician who was blinded to the study groups and at the initial visit, the women were familiarized with the location of the PFM and the pelvic anatomy and pathophysiology. After that information session, squeezing the PFM was shown in practice at least once to use in the urgency suppression strategies via digital palpation technique. In the second stage, including urgency suppression strategies, it was aimed to delay urination, to inhibit detrusor contraction and to prevent urgency; by squeezing the PFM several times in a row (women were encouraged to pause/stop their work, sit down if possible, relax the entire body and squeeze PFM repeatedly), breathing deeply, giving their attention to another job for a while and self-motivating (I can do it, I can check the urination, etc.). In the third stage, timed voiding program was started. It was carried out in 2 steps: timed voiding and increasing the time between urination considering the voiding diary. At the last stage, the women were encouraged to continue BT. By increasing their motivation that it is an effective treatment method, compliance to the treatment was increased.

Group 1: IVES (2 times in a week) This group included the IVES in addition to all components of the BT. IVES was performed in lithotomy position via electrical stimulation device with a vaginal probe. IVES sessions were performed two times in a week, for 10 weeks. Every session lasted 20 minutes. The intervention comprised a 20-sessions treatment program of ES. The stimulation parameters were frequency at 10 Hz, a 5-10s work-rest cycle and 100 ms pulse width. The symmetric biphasic pulse wave could be delivered over a range of 0-100 milliamp (mA). The intensity was controlled according to patients' discomfort level feedback.

Group 2: IVES (5 times in a week) This group also included the IVES in addition to all components of the BT as in Group 1. IVES performed in the same way as Group 1, except for frequency of treatment. IVES sessions were performed five times in a week, for 4 weeks. Every session lasted 20 minutes. The intervention comprised a 20-sessions treatment program of ES. Stimulation parameters were the same as Group 1.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 18 years old with clinical diagnosis of idiopathic overactive bladder
* Not tolerated or unresponsive to antimuscarinics and discontinued at least 4 weeks
* Able to give written, informed consent
* Able to understand the procedures, advantages and possible side effects
* Willing and able to complete the voiding diary and quality of life questionnaire
* The strength of pelvic floor muscle score 3/5 and more

Exclusion Criteria:

* Women with stress urinary incontinence
* History of conservative therapy for idiopathic overactive bladder within 6 months
* Pregnancy or intention to become pregnant during the study
* Current vulvovaginitis or urinary tract infections or malignancy
* History of urogynecological surgery within 3 months
* Anatomic structural disorders of genital region that could not allow to apply the vaginal probe
* More than stage 2 according to the pelvic organ prolapse quantification
* Cardiac pacemaker or implanted defibrillator
* Neurogenic bladder, signs of neurologic abnormalities at objective examination; history of the peripheral or central neurologic pathology
* Ultrasonographic evidence of post-void residual urine volume > 100 ml
* Allergy to condom or lubricant gel that is used with perineometer/vaginal probe

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women ≥ 18 years old with clinical diagnosis of idiopathic overactive bladder
Enrollment: 52 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Incontinence episodes-Incontinence related outcome measure | 20 minutes
  Women with a 50% or greater reduction in incontinence episodes were considered positive responders

SECONDARY OUTCOMES:
Severity of incontinence-Incontinence related outcome measure | 20 sessions (each sessions is 20 minutes )
  The 24-hour pad test was carried out to evaluate urinary loss
Nocturia-Incontinence related outcome measure | 20 sessions (each sessions is 20 minutes )
  It was used "nocturia" from data with a 3-day bladder diary
Frequency-Incontinence related outcome measure | 20 sessions (each sessions is 20 minutes )
  It was used "frequency" from data with a 3-day bladder diary
Number of Pads-Incontinence related outcome measure | 20 sessions (each sessions is 20 minutes )
  It was used "number of bads" from data with a 3-day bladder diary
Symptom severity-Incontinence related outcome measure | 20 sessions (each sessions is 20 minutes )
  Overactive Bladder Questionnaire (OAB-V8) was used to evaluate symptom severity in patients with in the study.
PFM strength-Incontinence related outcome measure | 20 sessions (each sessions is 20 minutes )
  To evaluate the PFM strength perineometer device
Quality of Life (QoL)-Incontinence related outcome measure | 20 sessions (each sessions is 20 minutes )
  The incontinence Impact Questionnaire (IIQ-7)scale was used to assess the patient's QoL associated with incontinence problem. The Scale has a minimum score of 0 and a maximum score of 21. Higher scores indicate worse incontinence related QoL.
Cure measured by 24-hour pad test | 20 sessions (each sessions is 20 minutes )
  In 24-hour pad test, incontinence that was under 1.3 gr was considered as a cure.
Improvement rate-Incontinence related outcome measure | 20 sessions (each sessions is 20 minutes )
  The improvement was assessed in terms of 50% and more reduction in wet weight compared to baseline measurements in the 24-hour pad test.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Kınıklı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No